CLINICAL TRIAL: NCT04686045
Title: Stroke Prevention in Atrial Fibrillation Patients Between 2004 and 2020
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jan Kochanowski University (Other)
Responsible Party: Principal Investigator, Iwona Gorczyca, MD PhD, Jan Kochanowski University
Other Study IDs: The Jan Kochanowski Uniwersity
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation; Stroke Prevention
MeSH Terms: conditions — Atrial Fibrillation | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
Prevention of thromboembolic complications is an important part in the management of patients with atrial fibrillation (AF). European and American guidelines recommend the use of non-vitamin K antagonist oral anticoagulants (NOACs) over therapy with vitamin K antagonists (VKA) in most AF patients. The number of patients treated with NOACs has increased significantly during the last few years. In the primary randomized controlled trials leading to their approval, compared to warfarin, NOACs were shown to be either noninferior or superior for stroke prevention in AF, with similar or reduced rates of bleeding, especially intracranial haemorrhage.

The aim of this study was to assess the frequency of oral anticoagulants using, espescially apixaban, dabigatran, and rivaroxaban, and the predictors of their prescription in a group of hospitalised patients with AF.

ELIGIBILITY:
Inclusion Criteria:

- non-valvular atrial fibrillation

Exclusion Criteria:

* valvular atrial fibrillation
* death during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with AF treated in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
oral anticoagulant treatment | one year

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - 1st Clinic of Cardiology and Electotherapy, Kielce, Grunwaldzka 45
  - Iwona Gorczyca, Kielce

IPD SHARING:
Plan to Share IPD: Undecided